CLINICAL TRIAL: NCT01146093
Title: Single Dose Two-Way Crossover Fed Bioequivalence Study of Pravastatin 80 mg Tablets in Healthy Volunteers
Brief Title: Bioequivalence Study of Pravastatin Sodium Tablets 80 mg Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Director, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AAI-US-138
Record Dates: First submitted 2010-02-10; First posted 2010-06-17 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
MeSH Terms: interventions — Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pravastatin Sodium Tablets 80 mg (Experimental): Dr.Reddy's Laboratories Limited
  Interventions: Drug: Pravastatin Sodium
- Pravachol 80 mg Tablets (Active Comparator): Bristol Myers Squibb
  Interventions: Drug: Pravastatin Sodium

INTERVENTIONS:
Drug: Pravastatin Sodium — Pravastatin Sodium Tablets 80 mg
  Other Names: Pravachol 80 mg tablets

SUMMARY:
This is a single Dose Two-Way Crossover Fed Bioequivalence Study of Pravastatin 80 mg Tablets of Dr.Reddy's Laboratories Limited with Pravachol 80mg, Bristol Myers Squibb in Healthy Volunteers.

DETAILED DESCRIPTION:
Single Dose Two-Way Crossover Fed Bioequivalence Study of Pravastatin 80 mg Tablets of Dr.Reddy's Laboratories Limited with Pravachol 80 mg, Bristol Myers Squibb in Healthy Volunteers.

A total of 24 non-smoking subjects (18 men and 6 women) were included in this study, of which 23 finished the study according to the protocol.

The washout period (7 days) between the two periods of the study and with an equal number of subjects randomly assigned

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females at least 18 years of age inclusive.
* Informed of the nature of the study and given written informed consent.
* Have a body weight within 15% of the appropriate range as defined in the 1983 Metropolitan Life Company tables and weighing at least 100 lbs. (Appendix I and II).

Exclusion Criteria:

* Hypersensitivity to Pravastatin (pravachol®), or similar compounds.
* Any history of a clinical condition which might affect drug absorption, metabolism or excretion.
* Recent history (within 1 year) of mental illness, drug addiction, drug abuse or alcoholism.
* Donation of greater than 500 m1 of blood in the past 4 weeks prior to study dosing or difficulty in donating blood.
* Received an investigational drug within the 4 weeks prior to study dosing.
* Currently taking any prescription medication, except oral contraceptives, within the 7 days prior to study dosing or over-the-counter medication within 3 days of study dosing. This prohibition does not include vitamins, or herbal preparations taken as nutritional supplements for non-therapeutic indications as judged by the attending physician.
* Tobacco use (>5 cigarettes per day) in the 3 months prior to study dosing.
* If female, the subject is lactating or has a positive pregnancy test at screening and prior to each of the two treatment periods. Females of child bearing potential must use a medically acceptable method of contraception throughout the entire study period and for one week after the study is completed. Medically acceptable methods of contraception that may be used by the subject and/or her partner are: oral contraceptives, progestin injection or implants, condom with spermicide, diaphragm with spermicide, IUD, vaginal spermicidal suppository, surgical sterilization of their partner(s) or abstinence. Females taking oral contraceptives must have taken them consistently for at least three months prior to receiving study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-11; Primary Completion 2002-11 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Scallion EE, MD, Principal Investigator — AAI, 6101 Quadrangle Drive, Chapel Hill, NC 27514